CLINICAL TRIAL: NCT05564351
Title: Evaluation of the Effect of Ear Plug and Eye Mask Use on Sleep Quality in Intensive Care patıents: Randomized Controlled Study
Brief Title: Ear Plug and Eye Mask Use on Sleep Quality in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, AYSUN KAZAK, Lecturer, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: "A.KAZAK33-H.TOPALI31"!
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Sleep Quality
Keywords: Nursing, intensive care unit, ear plug, eye mask, sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ear plug group (Experimental)
  Interventions: Other: eye mask and ear plug
- Eye mask group (Experimental)
  Interventions: Other: eye mask and ear plug
- Eye mask+Ear plug group (Experimental)
  Interventions: Other: eye mask and ear plug
- Control group (No Intervention)

INTERVENTIONS:
Other: eye mask and ear plug — black eye mask and silicon ear plug
  Arms: Ear plug group; Eye mask group; Eye mask+Ear plug group

SUMMARY:
This study was conducted as a pre-test and post-test randomized controlled single center study to evaluate the effect of ear plugs and eye mask application on sleep quality in patients hospitalized in the intensive care unit. 120 patients who received inpatient treatment in Siirt State Hospital general intensive care unit constitute the sample of the study. The sample consist of four groups: ear plug group (n=30), eye mask group (n=30), earplug-eye mask group (n=30) and control group (n=30). Data were collected using the "Patient Identification Form, Glasgow Coma Skale, Visual Analog Scale, Richards-Campbell Sleep Questionnaire (RCSQ), ear plug and eye mask". As a preliminary test, RCSQ was applied in the morning of the second day after the first night sleep of the patients. Then, according to the group they were assigned to, the patients were allowed to sleep by applying only ear plug, eye mask only and simultaneous ear plug-eye mask between 22:00-06:00. As a final test, RCSQ was readministered to patients on the morning of the third day after the second night's sleep. During the analysis of the data, frequency, number, mean, Student t test and/or Mann- Whitney U test, ANOVA and/or Kruskal- Wallis test, t test or Wilcoxon Sign test, chi-square test were used.

ELIGIBILITY:
Inclusion Criteria:

Being 18 years or older

* Being literate
* No hearing impairment
* Ability to communicate verbally
* Receiving inpatient treatment in the GICU for at least 3 days
* Have 15 Glasgow Coma Scale (GCS) scores (Minimum scores will be as follows. 3 points from eye response; 5 points from motor response; 2 points from verbal response)
* Agreeing to participate in the research

Exclusion Criteria:

Having a Visual Analog Scale (VAS) score above 7

* Using sleeping pills or sedative drugs
* Being treated with a diagnosis of sleep disorder
* Being on mechanical ventilation
* Having an active ear or eye infection
* Having a diagnosed psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Richards Campbell Sleep Scale | Three day
  RCSS is a six-item scale that evaluates the depth of night sleep, the time to fall asleep, the frequency of waking, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment.

SECONDARY OUTCOMES:
Visual Analog Scale | Three day
  The scale developed by Price et al. in 1983 measures the severity of the patient's pain.

OTHER OUTCOMES:
Glasgow Coma Scale | Three day
  The GCS was developed in Scotland/Glasgow in 1974 and is an international measurement tool that reflects the patient's state of consciousness. In the GCS, scoring is done in three separate sections: eye opening, verbal and motor response.
Patient Information Form | one day
  In this form, which was created by the researchers by scanning the literature; There are 13 questions in total, including patients' age, gender, marital status, education level, medical diagnosis, chronic diseases, drugs used, length of hospital stay and sleep habits, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Siirt State Hospital, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No